Project Title: Evaluation of Diagnostic Tools "Lateral Flow Immunoassay and FilmArray Warrior Panel" of Human Plague in Madagascar (Testing Multi-Echelon Diagnostics in a Resource Limited Endemic Setting: Human Plague in Madagascar)

**Document:** NAU ENG\_2020 Sign Consent\_CTR DOC DB#28.1

NCT Number: NCT04562012

Date Last Modified: 09APRIL2020

Project Number: 1582884-2 Expiration Date: April 19, 2021 This stamp must be on all consenting documents



## Annexe 3: Informed consent form

Project Title: « Evaluation of diagnostic tools (Lateral Flow Immunoassay and FilmArray Warrior Panel) of human plague in Madagascar » **Promoter**: Institut Pasteur de Madagascar-Plague Unit-Central Plague Laboratory I, the undersigned (last name, first name): Birthdate: Address: If it's a child, Name and surname of one of the parents / guardian ☐ Declares to have understood or to have explained to me the attached patient information leaflet on this study. I had the opportunity to ask any questions I wanted to the investigator (last name, first name):..... ☐ Accept freely and voluntarily to participate / that my child participates in this research of which the Pasteur Institute of Madagascar is responsible □ Accepts blood collection / on my child by a peripheral venous collection at the bend of the elbow and by finger prick. ☐ Give permission for my blood samples to be stored and used for further studies in Madagascar to better characterize the disease. □ I understand that the data concerning my child / myself, collected during this study, will remain STRICTLY CONFIDENTIAL and may only be consulted by the investigators and researchers involved in the project or, by persons mandated by the Pasteur Institute of Madagascar. All these people are subject to strict professional secrecy. ☐ I understand the investigators involved in the project (in Madagascar and abroad) can have access to the data from this study. ☐ I understand that Defense Threat Reduction Agency Broad (DTRA) via Northern Arizona University is the funding source. ☐ At the end of this study, I will be able to obtain the results of the biological analyzes carried out with the collected blood samples. Made in: Signature: the: